CLINICAL TRIAL: NCT03101293
Title: A Randomized, Open-Label, Single-Dose, 2-Period, Crossover Design, Phase 1 Study to Evaluate the Effect of Food on the Pharmacokinetics of TAK-831 T2 Tablet Formulation in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics of TAK-831 Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-831-1004; U1111-1189-8001 (Registry Identifier: WHO)
Record Dates: First submitted 2017-03-28; First posted 2017-04-05 (Actual); Results first posted 2019-03-18 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-831 400 mg Fasted + TAK-831 400 mg Fed (Experimental): TAK-831 400 mg, film-coated tablets, orally under fasted state, once on Day 1 of Intervention Period 1, followed by 7 days washout period, further followed by TAK-831 400 mg, film-coated tablets, orally under fed state, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-831
- TAK-831 400 mg Fed + TAK-831 400 mg Fasted (Experimental): TAK-831 400 mg, film-coated tablets, orally under fed state, once on Day 1 of Intervention Period 1, followed by 7 days washout period, further followed by TAK-831 400 mg, film-coated tablets, orally under fasted state, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-831

INTERVENTIONS:
Drug: TAK-831 — TAK-831 film-coated tablet.

SUMMARY:
The purpose of this study is to determine the pharmacokinetic (PK) of a single oral dose of TAK-831 400 milligram (mg) in the fasted state and to estimate the effect of food on the PK of a single oral dose of TAK-831 400 mg when administered as tablet formulation in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. TAK-831 is being tested in healthy participants under fasting and fed conditions in order to determine the effect of food on the PK of single oral dose of TAK-831 tablet formulation. The study will enroll approximately 16 participants. Participants will be randomly and equally assigned (by chance, like flipping a coin) to 1 of the 2 treatment sequences following as:

* TAK-831 400 mg Fasted + TAK-831 400 mg Fed
* TAK-831 400 mg Fed + TAK-831 400 mg Fasted All participants will be asked to take single oral dose of TAK-831 tablet at the same time on Day 1 of each Intervention Period. This single center trial will be conducted in the United States. The overall time to participate in this study is 23 days. Participants will visit the clinic on Day -1 and remained confined until Day 3 of Intervention Period 1 and 2. A washout period of minimum 7 days will be maintained between the doses in each Intervention Period. Participants will make 3 visits to the clinic on Days 4, 6 and 8 on each Intervention Period and will be contacted by telephone 14 days after the last dose of study drug (Day 23) for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs greater than or equal to (>=) 45 kilogram (kg) and has a body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.

Exclusion Criteria:

1. Has received TAK-831 in a previous clinical study.
2. Has poor peripheral venous access.
3. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to first dose of study drug.
4. Has any dietary restrictions or preferences that may interfere with the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 04 April 2017 to 26 May 2017.
Pre-assignment Details: Healthy participants were enrolled in this 2-way crossover study and randomized in 1 of the 2 treatment sequences which determined the order to receive TAK-831 400 milligram (mg) film-coated tablets under fasted conditions and TAK-831 400 mg tablet under fed conditions (nutritional drink).
Groups:
- TAK-831 400 mg Fasted + TAK-831 400 mg Fed: TAK-831 400 mg, film-coated tablets, orally, under fasted state, once on Day 1 of Intervention Period 1, followed by at least 7 days of washout period, further followed by TAK-831 400 mg, tablet, orally, under fed state, once on Day 1 of Intervention Period 2.
- TAK-831 400 mg Fed + TAK-831 400 mg Fasted: TAK-831 400 mg, film-coated tablets, orally, under fed state, once on Day 1 of Intervention Period 1, followed by at least 7 days of washout period, further followed by TAK-831 400 mg, tablet, orally, under fasted state, once on Day 1 of Intervention Period 2.
Period: Intervention Period 1
Arm/Group | TAK-831 400 mg Fasted + TAK-831 400 mg Fed | TAK-831 400 mg Fed + TAK-831 400 mg Fasted
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | TAK-831 400 mg Fasted + TAK-831 400 mg Fed | TAK-831 400 mg Fed + TAK-831 400 mg Fasted
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0
Not completed — Positive drug urine screen | 1 | 0
Period: Intervention Period 2
Arm/Group | TAK-831 400 mg Fasted + TAK-831 400 mg Fed | TAK-831 400 mg Fed + TAK-831 400 mg Fasted
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-831 400 mg Fasted + TAK-831 400 mg Fed | TAK-831 400 mg Fed + TAK-831 400 mg Fasted | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  years | 35.4 (7.98) | 32.6 (11.22) | 33.9 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Female | 1 | 2 | 3
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 6 | 8 | 14
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 3 | 6
    White | 3 | 5 | 8
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    United States | 7 | 8 | 15
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  kilogram (kg) | 73.3 (9.65) | 78.6 (11.19) | 76.1 (10.48)
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  centimeter (cm) | 171.3 (6.40) | 173.8 (7.19) | 172.6 (6.71)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  kilogram per square meter (kg/m^2) | 24.9 (2.17) | 25.9 (2.45) | 25.5 (2.30)
Smoking Classification [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Never smoked | 5 | 7 | 12
    Current smoker | 1 | 0 | 1
    Ex-smoker | 1 | 1 | 2
Alcohol Classification [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Never drunk | 3 | 3 | 6
    Current drinker | 4 | 5 | 9
    Ex-drinker | 0 | 0 | 0
Caffeine Consumption [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Caffeine consumption | 6 | 7 | 13
    No caffeine consumption | 1 | 1 | 2
Xanthine Consumption [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Xanthine consumption | 6 | 7 | 13
    No xanthine consumption | 1 | 1 | 2
Female Reproductive Status [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Post-menopausal | 0 | 1 | 1
    Surgically sterile | 1 | 1 | 2
    Not applicable (Male) | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-831 400 mg Fasted: TAK-831 400 mg, film-coated tablets, orally, under fasted state, once on Day 1 of either Intervention Period 1 or Intervention Period 2.
- TAK-831 400 mg Fed: TAK-831 400 mg, film-coated tablets, orally, under fed state, once on Day 1 of Intervention Period 1 or Intervention Period 2.
Arm/Group | TAK-831 400 mg Fasted | TAK-831 400 mg Fed
Number analyzed (Participants) | 15 | 14
nanogram per milliliter (ng/mL) | 650.04 (47.7) | 865.48 (53.5)
Statistical Analysis 1: Comparison: TAK-831 400 mg Fasted vs TAK-831 400 mg Fed; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as fixed effects and participant nested within sequence as a random effect. The least squares means and difference of least squares means for the log-transformed parameters were exponentiated to obtain the point estimates of the food effect and 90% confidence intervals (CIs); p = 0.0058, ANOVA; LS Mean Ratio = 1.343, 90% CI 2-sided [1.146 to 1.574]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-831 400 mg Fasted | TAK-831 400 mg Fed
Number analyzed (Participants) | 15 | 14
hour*nanogram per milliliter (h*ng/mL) | 2290.8 (53.1) | 2535.6 (58.8)
Statistical Analysis 1: Comparison: TAK-831 400 mg Fasted vs TAK-831 400 mg Fed; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as fixed effects and participant nested within sequence as a random effect. The least squares means and difference of least squares means for the log-transformed parameters were exponentiated to obtain the point estimates of the food effect and 90% CIs; p = 0.1763, ANOVA; LS Mean Ratio = 1.121, 90% CI 2-sided [0.969 to 1.298]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration. The PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-831 400 mg Fasted | TAK-831 400 mg Fed
Number analyzed (Participants) | 13 | 10
h*ng/mL | 2194.8 (53.1) | 2465.9 (67.8)
Statistical Analysis 1: Comparison: TAK-831 400 mg Fasted vs TAK-831 400 mg Fed; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.2745, ANOVA; LS Mean Ratio = 1.154, 90% CI 2-sided [0.929 to 1.433]

4. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Treatment-emergent Adverse Event (TEAE)
Time Frame: Day 1
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-831 400 mg Fasted | TAK-831 400 mg Fed
Number analyzed (Participants) | 15 | 14
percentage of participants | 0 | 7.1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 14 days after the last dose of study drug (up to Day 23)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-831 400 mg Fasted | TAK-831 400 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAK-831 400 mg Fasted (N=15) | TAK-831 400 mg Fed (N=14)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03101293/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03101293/SAP_001.pdf